CLINICAL TRIAL: NCT05846204
Title: The Effect of Progressive Muscle Relaxation and Deep Breathing Exercises Training on Dyspnea, Fatigue and, Quality of Sleep in Patients With COPD: A Randomized Controlled Clinical Trial
Brief Title: Progressive Muscle Relaxation and Deep Breathing Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, NİHAN TÜRKOĞLU, Assist Prof., Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AtaturkUnıv
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Progressive Muscle Relaxation; Deep Breath; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PMR Group (Experimental): The PMR exercise, which includes the systematic relaxation of the main muscle groups of the body aimed at physical and psychological relaxation, was applied twice a day, every weekday, for eight weeks. PMR exercises and training on the application of these exercises were given to the patients individually by face-to-face interview method. During the training process, "Muscle Relaxation Exercises Practice Guide" and "Relaxation Exercises Audio Recordings", which were prepared by the researcher and included relaxation exercises, were used. Voice recordings were uploaded to each patient's mobile phone so that they could continue the application at home. The steps of the relaxation exercises were explained to the patient by the researcher and he was shown exactly how to do the exercises.
  Interventions: Behavioral: Progressive Muscle Relaxation
- Deep Breath Group (Experimental): WB exercises training was given to the patients in this group individually by face-to-face interview. During the application, the importance of deep and comfortable breathing was explained and correct breathing technique was taught. Informing and application training took an average of 20-25 minutes for each patient. The patients were told to do the 10-minute application at home 3 times a day for 8 weeks. They were called once a week and asked whether they continued the practice and whether they had any difficulties during the exercises.
  Interventions: Behavioral: Deep Breathing Exercise Group-DBE
- Control (No Intervention): No intervention will be applied to the control group.

INTERVENTIONS:
Behavioral: Progressive Muscle Relaxation — The PMR exercise, which includes the systematic relaxation of the main muscle groups of the body aimed at physical and psychological relaxation, was applied twice a day, every weekday, for eight weeks.
  DB exercises training was given to the patients in this group individually by face-to-face interview. During the application, the importance of deep and comfortable breathing was explained and correct breathing technique was taught.
  Arms: PMR Group
Behavioral: Deep Breathing Exercise Group-DBE — Breathing exercise is an exercise to improve breathing and functional performance. deep breathing exercise; It is a nursing intervention that helps to increase the function of respiratory muscles and improve ventilation and oxygenation.
  Arms: Deep Breath Group

SUMMARY:
The population of the study was composed of 186 patients whose cells were assigned to Atatürk University Hospital Educational Diseases Polyclinic between April and June 2023, and whose cells were found to have COPD according to the Chronic Obstructive Pulmonary Disease Initiative by the physician. A total of 140 patients approved the inclusion criteria and agreed to participate in the study. Priori power analysis was performed for sampling determination. In the power analysis, Cohen's medium effect size reference method was chosen. As a result of the power analysis, it was determined that it should be done with a total of 90 patients, 30 patients in each group, two experimental groups and the control group (α=0.05, power=0.8, and effect expectation=0.65). In case of data loss, this number plus approximately 20% reserve allocation included 36 patients in each group. However, the study was completed with a total of 96 patients, including PMR(n=31), DB(n=32) and 33 control subjects.

DETAILED DESCRIPTION:
The PMR exercise, which includes the systematic relaxation of the main muscle groups of the body aimed at physical and psychological relaxation, was applied twice a day, every weekday, for eight weeks. PMR exercises and these exercises were given to the patients individually.

The training for the implementation of the exercises was given by face-to-face interview method. During the training process, "Muscle Relaxation Exercises Practice Guide" and "Relaxation Exercises Audio Recordings", which were prepared by the researcher and included relaxation exercises, were used.

Deep Breath exercises training was given to the patients in this group individually by face-to-face interview. During the application, the importance of deep and comfortable breathing was explained and correct breathing technique was taught. Informing and application training took an average of 20-25 minutes for each patient. The patients were told to do the 10-minute application at home 3 times a day for 8 weeks. They were called once a week and asked whether they continued the practice and whether they had any difficulties during the exercises.

ELIGIBILITY:
Inclusion Criteria:

* Not having any physical problems
* Conscious
* Fully oriented
* Not have an acute exacerbation attack in the past month

Exclusion Criteria:

* Having a hearing problem,
* Inability to practice relaxation exercises regularly,
* Wanting to leave the study
* Neurological diseases,
* Those with comorbidities such as acute myocardial infarction or cancer,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Chronic Obstructive Pulmonary Disease and Asthma Fatigue Scale | two week
  The COPD and Asthma Fatigue Scale (CAFS) was developed by Revicki et al. In the scale consisting of a total of 12 questions, the items of the questions are graded in a Likert type. The total raw score is obtained by summing all item scores, and the raw scores are converted to a total scale score between 0 and 100 points. The increase in the scale score indicates the increase in the fatigue level of the person.
Dyspnea-12 Scale | Two week
  The scale developed by Yorke et al. consists of 12 items measuring the severity of dyspnea. It consists of 4-point Likert type options. The highest score that can be obtained from the physical sub-dimension of the scale is 21, and the highest score that can be obtained from the emotional sub-dimension is 15. The lowest score of the scale is 0, and the highest score is 36. An increase in the score obtained from the scale indicates an increase in the severity of dyspnea.
Pittsburgh Sleep Quality Index | Two week
  Designed by PSQI, Buysee et al. PSQI specifically measures subjective sleep quality over a one-month period. The PSQI includes 19 items on seven subscales: subjective sleep quality, sleep duration, sleep disturbance, sleep delay, sleep efficiency, use of sleep medication, and daytime dysfunction. Items are scored on a 4-point Likert scale from 0 to 3 points. Scores of the subscales are added to an overall PSQI score. The total score of the questionnaire ranges from 1 to 21 points, where scores higher than 5 indicate poor sleep quality and scores lower than 5 indicate no sleep disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: Nihan Türkoğlu, Assist.Prof., Study Chair — Ataturk University
Locations (1):
- Ataturk Unıversity, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No